CLINICAL TRIAL: NCT04417777
Title: Etude génétique Des Dilatations Des Bronches Idiopathiques en Polynésie française
Brief Title: Genetic Study of the Dilatations of the Idiopathic Bronchi in French Polynesia
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: POLYGENET
Record Dates: First submitted 2020-05-26; First posted 2020-06-05 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Bronchiectasis
Keywords: Genetic Disease; Idiopathic Bronchiectasis Polynesia; polynesia
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ADN and ARN are collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polynesian patient: Patient with dilatation of idiopathic bronchi
  Interventions: Genetic: Blood Test
- Relatives of polynesian patient: Healthy
  Interventions: Genetic: Blood Test

INTERVENTIONS:
Genetic: Blood Test — Blood analysis

SUMMARY:
Bronchiectasis, defined by an increase in bronchial caliber and thickening of the bronchial wall, is associated with recurrent respiratory infections, chronic cough and bronchorrhea, and a frequent progression to chronic respiratory failure. Investigator distinguish focal bronchiectasis usually resulting from a localized cause and diffuse bronchiectasis which the possible causes are multiple (immune deficiencies, genetic diseases, auto immune pathologies, aspergillosis broncho -allergic lung, sequelae of pulmonary infections).The etiological assessment is negative in 26 to 53% of cases, defining the idiopathic bronchiectasis. However, the discovery of an underlying cause can change the patient's management (up to 37% of cases).

Despite the lack of epidemiological data in French Polynesia, Australian and New Zealand studies found a high prevalence of bronchiectasis in Polynesians. Few clinical studies published in the early 1980s suggested a ciliary origin.

Due to its geographic characteristics, the Polynesian population constitutes an interesting ethnic group. Indeed, there is a low genetic mixing and the prevalence of certain genetic diseases like the syndrome of Alport or some hereditary retinal dystrophies are high. This type of population is very suitable for discovering new genes in human pathology.

Investigator decided to conduct an observational study to find an underlying genetic cause of bronchiectasis in Polynesians by performing a whole exome sequencing. Investigator chose to study index cases defined by an upset of symptoms during the childhood, a family history of idiopathic bronchiectasis, and/or a consanguinity. Investigator also want to study healthy first degree relatives, in order to be able to better identify the clinical significant of DNA variants and focus the analysis on those that may be pathogenic

ELIGIBILITY:
*Patients

Inclusion Criteria:

* Polynesian adult more than18 years
* dilatation of idiopathic bronchi confirmed to thoracic CTscan
* Negative etiological balance (including sweat test, research of Dyskinesia Ciliary Primitive and immunological check-up)
* Appearance of symptoms in childhood, or family history of chronic bronchial disease, or notion of inbreeding
* Signed consent
* Affiliated with a social security system

Exclusion Criteria:

* Refusal to participate in the study

  *Relatives
* First-degree healthy relatives
* Polynesian adult more than 18 years
* Signed consent
* Affiliated with a social security system

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Polynesian patient with dilatation of idiopathic bronchi
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
identification of genetic mutation | Anytime in the period of 10 years
  New mutation in the coding region or mutation located outside the coding regions on the transcriptome

SECONDARY OUTCOMES:
Clinical phenotype | Anytime in the period of 10 years
  Extra-respiratory history Bronchial colonizations Scannographic aspect
scannographic description | Anytime in the period of 10 years
  Extra-respiratory history Bronchial colonizations Scannographic aspect
Effect on the splicing of messenger RNA | Anytime in the period of 10 years
  correlation genotype/phenotype
transcriptome of patients | Anytime in the period of 10 years
  correlation genotype/phenotype

CONTACTS AND LOCATIONS:
Locations (1):
- CH Polynesie Française, Papeete, French Polynesia